CLINICAL TRIAL: NCT02726932
Title: Intra-abdominal View and Inflammatory Markers in Secondary Peritonitis - Correlation to Recovery
Acronym: PERICLASS
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Matti Tolonen, M.D., Helsinki University Central Hospital
Other Study IDs: Dnro 6/13/03/02/2016
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Peritonitis
Keywords: Peritonitis; Inflammatory Markers; Patient Outcome Assessment; Classification; Multiple Organ Failure; Intraabdominal Infections
MeSH Terms: conditions — Peritonitis; Multiple Organ Failure; Intraabdominal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — Whole blood sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention, merely observational

SUMMARY:
The purpose of this study is to analyze the correlation between intra-abdominal view and patient recovery in secondary peritonitis, and to create a new classification based on these results. Additionally, a variety of inflammatory markers from blood samples will be collected in order to analyze their correlation with patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients > 18 years old
* operated for complicated intra-abdominal infection

Exclusion Criteria:

* another diagnosis requiring ICU level care at the same time
* acute pancreatitis
* acute mesenteric ischaemia due to occlusion in superior mesenteric artery or vein
* peritonitis due to timely diagnosed trauma
* missing informed consent or inability to understand it

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients operated for complicated intra-abdominal infection in a single university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days
  Death within 90 days of primary operation for diffuse peritonitis
ICU admission | 90 days
  Intensive Care Unit admission and length of ICU treatment
Length of hospitalization | 90 days
  Days in hospital postoperatively
Reoperations | 90 days
  Reoperations needed postoperatively
Complications | 90 days
  Postoperative complications according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Panu Mentula, M.D., Ph.D., Study Chair — Helsinki University Central Hospital, Abdominal Center, Gastrointestinal Surgery
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tolonen M, Sallinen V, Leppaniemi A, Backlund M, Mentula P. The role of the intra-abdominal view in complicated intra-abdominal infections. World J Emerg Surg. 2019 Mar 29;14:15. doi: 10.1186/s13017-019-0232-7. eCollection 2019. PMID 30976292